CLINICAL TRIAL: NCT06384911
Title: InvesT1D: Promoting Adolescent Investment in Diabetes Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Davene R. Wright, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004543
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (low-value incentive, 6 months [24 weeks]) (Experimental): If the participant is assigned to Group A, they would receive $1.75 for each day that they meet their diabetes self-management goal. This equates to up to $49 every 4 weeks ($1.75 x 28 days = $49), or up to $294 over a period of 24 weeks. They would also receive $2.75 for each week that they meet their clinical outcome goal. This equates to up to $11 every 4 weeks ($2.75 x 4 weeks), or up to $66 over a period of 24 weeks. In total, they could earn up to $60 ($49 + $11) every 4 weeks, or up to $360 over a period of 24 weeks.
  Interventions: Behavioral: Financial Incentives Program
- Group B (high-value incentive, 6 months [24 weeks]) (Experimental): If the participant is assigned to Group B, they would receive $3.50 for each day that they meet their diabetes self-management goal. This equates to up to $98 every 4 weeks ($3.50 x 28 days = $98), or up to $588 over a period of 24 weeks. They would also receive $5.50 for each week that they meet their clinical outcome goal. This equates to up to $22 every 4 weeks ($5.50 x 4 weeks), or up to $132 over a period of 24 weeks. In total, they could earn up to $120 ($98 + $22) every 4 weeks, or up to $720 over a period of 24 weeks.
  Interventions: Behavioral: Financial Incentives Program
- Group C (low-value incentive, 12 months [48 weeks]) (Experimental): If the participant is assigned to Group C, they would receive $1.75 for each day that they meet their diabetes self-management goal. This equates to up to $49 every 4 weeks ($1.75 x 28 days = $49), or up to $588 over a period of 48 weeks. They would also receive $2.75 for each week that they meet their clinical outcome goal. This equates to up to $11 every 4 weeks ($2.75 x 4 weeks), or up to $132 over a period of 48 weeks. In total, they could earn up to $60 ($49 + $11) every 4 weeks, or up to $720 over a period of 48 weeks.
  Interventions: Behavioral: Financial Incentives Program
- Group D (high-value incentive, 12 months [48 weeks]) (Experimental): If the participant is assigned to Group C, they would receive $1.75 for each day that they meet their diabetes self-management goal. This equates to up to $49 every 4 weeks ($1.75 x 28 days = $49), or up to $588 over a period of 48 weeks. They would also receive $2.75 for each week that they meet their clinical outcome goal. This equates to up to $11 every 4 weeks ($2.75 x 4 weeks), or up to $132 over a period of 48 weeks. In total, they could earn up to $60 ($49 + $11) every 4 weeks, or up to $720 over a period of 48 weeks.
  Interventions: Behavioral: Financial Incentives Program
- Group E (usual care, 6 months [24 weeks]) (No Intervention): Usual care reflects the standard treatment currently provided to adolescents with type 1 diabetes at Seattle Children's Hospital. All adolescent participants in the study will have access to the multidisciplinary care team including a diabetes provider, registered diabetes nurse, social worker, and nutritionist. They will continue to be offered routine diabetes clinic appointments as is the standard of care. Telephone consultations are available 24/7 as often as necessary between clinic visits.
- Group F (usual care, 12 months [48 weeks]) (No Intervention): Usual care reflects the standard treatment currently provided to adolescents with type 1 diabetes at Seattle Children's Hospital. All adolescent participants in the study will have access to the multidisciplinary care team including a diabetes provider, registered diabetes nurse, social worker, and nutritionist. They will continue to be offered routine diabetes clinic appointments as is the standard of care. Telephone consultations are available 24/7 as often as necessary between clinic visits.

INTERVENTIONS:
Behavioral: Financial Incentives Program — Adolescent participants will receive financial incentives for meeting diabetes self-management and clinical outcome goals.
  Arms: Group A (low-value incentive, 6 months [24 weeks]); Group B (high-value incentive, 6 months [24 weeks]); Group C (low-value incentive, 12 months [48 weeks]); Group D (high-value incentive, 12 months [48 weeks])

SUMMARY:
The goal of this clinical trial is to see if a financial incentives program called InvesT1D is helpful to support diabetes management in adolescents with type 1 diabetes.

Adolescent participants will be randomized to usual care or receive financial incentives for meeting diabetes self-management and clinical outcomes goals during the study. Researchers will compare changes in glucose levels, as well as adolescent and caregiver person-reported outcomes between groups.

DETAILED DESCRIPTION:
Adolescents face many challenges as they transition from childhood to adulthood. For adolescents with type 1 diabetes, there are additional responsibilities that come with daily diabetes self-management.

The goal of this study is to find out whether financial incentives can help adolescents with their daily self-management. Adolescent participants will be assigned to one of 6 groups. Some participants will be asked to choose diabetes self-management goals such as increasing daily bolus insulin administration or increasing their continuous glucose monitoring system wear time, and then will be provided with financial incentives (money) when they meet their selected goals. Other participants will be asked to continue their diabetes management as usual.

Researchers will collect data from 96 adolescent participants and their caregivers to assess change in glucose levels, as well as adolescent and caregiver person-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes ≥12 months
* Utilize a continuous glucose monitor (CGM) to support diabetes management
* Average daily CGM use is less than or equal to 70% of the time and/or their baseline average insulin bolus administration is less than or equal to 3 times a day
* Are using diabetes technology that allows for tracking of bolus insulin administration if participant wants to work on improving daily bolus insulin administration
* Cognitively able to participate in incentive program and complete surveys
* Have access to a mobile phone to receive information about goal attainment and incentive updates
* Have the ability to upload glucose and insulin administration data remotely per processes used by participant's diabetes care team
* Caregivers are willing to participate in study and complete surveys

Exclusion Criteria:

* At time of screening, average CGM wear is greater than 70% of the time or baseline average insulin bolus administration is greater than 3 times a day
* Adolescent is not interested in using diabetes technology that allows for tracking of bolus insulin administration if participant wants to work on improving daily bolus insulin administration
* Cognitively or physically unable to participate
* Adolescent is a ward of the state
* Severe comorbidities including other major chronic health conditions that significantly impact daily management demands or health outcomes
* Caregivers are not willing to participate in study and complete surveys

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Time In Range | Change over 12-18 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are in range (70-180 mg/dL)

SECONDARY OUTCOMES:
Time Above Range | Change over 12-18 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are above range (>180 mg/dL).
Time Below Range | Change over 12-18 months
  Continuous glucose monitor sensor glucose measurements collected during the intervention that are below range (<70 mg/dL).
Hemoglobin A1c (HbA1c) | Change over 12-18 months
  HbA1c laboratory measurements collected during the intervention.
Diabetes Distress | Change over 12-18 months
  Diabetes distress will be assessed with the Problem Areas in Diabetes Scale -- Teen Version. Higher scores indicate higher diabetes distress (scale: 14-84).
Diabetes Family Conflict | Change over 12-18 months
  Diabetes family conflict will be assessed with the Diabetes Family Conflict Scale. Higher scores indicate higher diabetes family conflict (scale: 19-57).
Adolescent Quality of Life | Change over 12-18 months
  Adolescent health-related quality of life will be assessed with the EQ-5D instrument. High score indicated higher health status (scale: 0-100).
Caregiver Quality of Life | Change over 12-18 months
  Caregiver quality of life will be assessed using the Care-related Quality of Life instrument. Higher scores represent higher caregiving burden (score: 0-100).
Diabetic Ketoacidosis | 12-18 months
  Episodes of severe hypoglycemia requiring emergency department visit or hospital admission will be extracted from medical record data.
Severe Hypoglycemia | 12-18 months
  Episodes of severe hypoglycemia requiring emergency department visit or hospital admission will be extracted from medical record data.
Insulin Adminstration | Change over 12-18 months
  Daily bolus insulin administration will be assessed based on data collected on insulin pump or inPen diabetes data management platforms.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The Harvard Dataverse repository provides searchable study-level metadata for dataset discovery. The repository assigns DOIs as persistent identifiers and has a robust preservation plan to ensure long-term access. Data will be discoverable online through standard web search of the study-level metadata as well as the persistent pointer from the DOI to the dataset. The dataset will be tagged with the NIH award number to facilitate searches.
Supporting Information: SAP
Time Frame: Data requests can be submitted at the end of the funding period and the data will be made accessible for up to 10 years.
Access Criteria: The Harvard Dataverse repository, is an open-source web application that provides searchable study-level metadata for dataset discovery. The repository assigns DOIs as persistent identifiers and has a robust preservation plan to ensure long-term access. Data will be discoverable online through standard web search of the study-level metadata as well as the persistent pointer from the DOI to the dataset. The dataset will be tagged with the NIH award number to facilitate searches.